CLINICAL TRIAL: NCT00263640
Title: A Multicentre Randomised Placebo-controlled Double-blind Clinical Trial for Evaluation of Safety and Efficacy of Specific Immunotherapy With an Alum.-Adsorbed Allergoid Preparation of House Dust Mite (D. Pteronyssinus) in Patients With Allergic Bronchial Asthma, Rhinitis, Rhinoconjunctivitis
Brief Title: Safety and Efficacy of House Dust Mite Allergoid in the Treatment of Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Al0104av; 2004-003892-35 (EudraCT Number)
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Hypersensitivity
Keywords: House dust mite; Bronchial Asthma; Allergy; House Dust Mite Allergy
MeSH Terms: conditions — Respiratory Hypersensitivity; Asthma; Hypersensitivity; Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo was given the same way as a subcutaneous (just under the skin) injection. Children received lifestyle counselling.
  Interventions: Drug: Placebo
- Acaroid (Experimental): The drug tested in this study (aluminium hydroxide-adsorbed house dust mite (D. pteronyssinus) allergoid preparation) was given as a subcutaneous injections of increasing doses.
  Interventions: Biological: Acaroid

INTERVENTIONS:
Biological: Acaroid — The drug tested in this study (aluminium hydroxide-adsorbed house dust mite (D. pteronyssinus) allergoid preparation) was given as a subcutaneous injections of increasing doses.
  Other Names: Specific Immunotherapy
  Arms: Acaroid
Drug: Placebo — Placebo was given the same way as a subcutaneous (just under the skin) injection. Patients were treated according the same dosing schedule of active group. Children received lifestyle counselling.
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
The trial is performed to assess efficacy and safety of the Allergopharma house dust mite allergoid in bronchial asthma.

DETAILED DESCRIPTION:
The rationale for the present study was to demonstrate clinical efficacy and tolerability compared to placebo in a phase III clinical study of pivotal character with a representative number of patients suffering from fully reversible asthma +/- allergic rhinitis. This condition is present in paediatric and adult patients with a shorter history of GINA II and III asthma, who were investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Bronchial asthma
* Requirements for inhaled corticosteroid
* Positive skin prick test to house dust mite
* Positive radioallergosorbent test (RAST) to house dust mite
* Positive provocation test result to house dust mite

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2005-05; Primary Completion 2009-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Inhalative dose of fluticasone propionate | After 2 years
  The primary endpoint variate was the change of inhalative dose of fluticasone propionate needed to ensure asthma control according to GINA recommendation.

SECONDARY OUTCOMES:
Pre-bronchodilator morning peak flow | After 2 years
  Post treatment, the changes from baseline in the mean pre-bronchodilator morning peak flow during the last two weeks of the diary phases were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator — Allergopharma GmbH & Co. KG
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- [Result] Zielen S, Kardos P, Madonini E. Steroid-sparing effects with allergen-specific immunotherapy in children with asthma: a randomized controlled trial. J Allergy Clin Immunol. 2010 Nov;126(5):942-9. doi: 10.1016/j.jaci.2010.06.002. Epub 2010 Jul 10. PMID 20624650
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de